CLINICAL TRIAL: NCT03304652
Title: Cerebral MRI During Sleep
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David Dubowitz, Associate Professor, University of California, San Diego
Other Study IDs: 170804
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Sleep
MeSH Terms: interventions — zaleplon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Zaleplon — Sleep Aid; 10mg; Oral; Single Use
  Other Names: Sonata
Other: Natural Sleep — Natural Sleep without medication

SUMMARY:
Recent studies in animal models have suggested a critical role for cerebrospinal fluid and Interstitial fluid flux through cerebral parenchyma for removal of byproducts of cellular metabolism and hence in maintaining the health of the brain. This effect is modulated during sleep, suggesting a potentially important mechanism for sleep to maintain both acute homeostasis and long-term cerebral health.

The central goal of these studies is to develop a sensitive MRI biomarker of cerebral conformational changes during sleep. This exploratory work aims to establish the sensitivity and reproducibility of MRI as a non-invasive neuroimaging assessment of cerebral changes during natural sleep and sedation.

DETAILED DESCRIPTION:
Recent studies in animal models have suggested a critical role for cerebrospinal fluid (CSF) / Interstitial fluid (ISF) flux through cerebral parenchyma for removal of byproducts of cellular metabolism and hence in maintaining the health of the brain. It remains unknown to what extent these phenomena exist in the human brain. A key challenge in this work is to make non-invasive and reproducible measurements of the cerebral microenvironment in humans. For these studies, the investigators have implemented a suite of MRI measurements to track physiological changes in the brain during sleep. This exploratory work aims to establish the sensitivity and reproducibility of MRI as a non-invasive neuroimaging assessment of cerebral changes during natural sleep and sedation. The long term goal of this work is to use MRI as an imaging biomarker to assess the cerebral response to normal versus disordered sleep in patients.

Our specific aims will address the following questions:

Aim 1: How sensitive are MRI metrics for determining changes in the brain during sleep?

Aim 2: How reproducible are MRI metrics during sleep and during sedation?

The investigators will recruit 12 normal adult subjects for this study (consecutive respondees to recruitment adverts). The investigators will make regional MRI measurements during onset, maintenance and waking from stage N2 sleep. From these the investigators will characterize which MRI metrics are most sensitive to changes in the cerebral environment, and how these vary for different cerebral regions.

Measurements will be repeated during ~90 minutes of natural sleep, and following oral sedation with 10 mg zaleplon (Sonata).

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults

Exclusion Criteria:

1. age not in range 18-59
2. smoking / recreational drug use
3. pregnant women / breast feeding
4. contraindication to MRI
5. contraindications to Zaleplon
6. history of cardiovascular pulmonary or cerebral disease (hypertension (diastolic >90 mmHg, systolic > 150 mmHg), unstable cerebrovascular syndromes, prior history of cardiac arrhythmias, unstable angina, chronic obstructive pulmonary disease).
7. Current SSRI antidepressant medication
8. History of sleep disorder or currently taking sedative / stimulant medication

Ages: 18 Years to 59 Years | Sex: All
Age Groups: Adult
Study Population: 12 normal adults for this study aged 18-59. Both male and female. Consecutive participant sampling
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Cerebral MRI Changes | 90 Minutes of Sleep
  Change in MRI Signal from Awake Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No